CLINICAL TRIAL: NCT07403799
Title: Real-life, Observational Study on Opicapone in Patients With Parkinson's Disease and Early Motor Fluctuations in Italy
Brief Title: REal-life ON PARKinson's - ITaly (REONPARK-IT)
Status: Recruiting | Type: Observational
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: IT-BIAL-9-402
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
Keywords: REONPARK-IT; Opicapone
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: To evaluate the long-term effectiveness of opicapone in patients with Parkinson's disease (PD) and early motor fluctuations by means of the Patient Global Impression of Change (PGI-C) at 12 months after start of treatment
  Interventions: Drug: Opicapone 50 mg

INTERVENTIONS:
Drug: Opicapone 50 mg — The recommended dose of opicapone is 50 mg. Opicapone must be taken once a day before going to bed, at least one hour before or one hour after levodopa combinations. As opicapone enhances the effects of levodopa, it could be necessary to adjust levodopa dose by extending the dosing intervals and/or reducing the amount of levodopa per dose within the first days to first weeks after initiating treatment with opicapone.

SUMMARY:
The present study aims to evaluate the effectiveness and safety of opicapone in a real-world setting at centers for Parkinson's disease located in Italy.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational cohort study of patients with Parkinson's Disease and early motor fluctuations treated with opicapone in Italy.

Treatment with opicapone will be independent from participation in this observational study and must not be initiated for the purpose of participating in it. Opicapone will be administered according to the local Summary of Product Characteristics (SmPC).

Data on patients will be collected in accordance with routine clinical visits and examinations starting from the date when patient consent is obtained, and for up to two years after start of treatment with opicapone. The collection of the patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO) will be dictated by the routine clinical practice at each center; thus, scales left blank will not be considered protocol deviations.

Patients will be followed up for a maximum of 2 years (±2 months). Because of the observational design of the study, there are no imposed visits beyond those performed as per clinical practice. Visits are however planned closest to 6 months (±2 months), 12 months (±2 months), 18 months (±2 months), and 24 months (±2 months) after inclusion.

The overall duration of the study will be of approximately 5 years, with 24 months of recruitment and 24 months (±2 months) of follow-up from the last patient in. The End of Study (EOS) is defined as the time when the last enrolled patient has completed 24 months (±2 months) of assessments (unless early termination) after enrolment.

In the event that a patient discontinues opicapone, he/she will be discontinued from the study. Patients discontinued from the study will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is able to comprehend and willing to provide written informed consent to participate in this study.
2. Patients aged 30 years or older.
3. The patient has a clinical diagnosis of PD according to the diagnostic criteria of United Kingdom (UK) PD Society Brain Bank (2006) or Movement Disorder Society (MDS) Clinical Criteria (2015).
4. Disease severity stages I-III (Hoehn & Yahr Staging).
5. The patient is on treatment with levodopa/DOPA decarboxylase inhibitors (DDCI) for at least 1 year.
6. The patient has signs of wearing off phenomenon/end-of dose motor fluctuations for less than 2 years.
7. Patients starting treatment with opicapone as per local Summary of Product Characteristics (SmPC). Initiation of treatment with opicapone will be independent from participation in this observational study and must not be initiated for the purpose of study participation. The decision to treat patients with opicapone will occur before patients are enrolled in the study.

Exclusion Criteria:

1. The patient has any form of Parkinsonism other than PD.
2. The patient is participating in a clinical trial with an investigational drug or has concluded participation within 30 days.
3. The patient has any contraindication to opicapone according to SmPC.
4. The patient meets criteria for dementia in the Investigator's judgment.
5. The patient is currently treated with catechol-O-methyl transferase (COMT) inhibitors.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at approximately 20 centers located in Italy and plans to enroll approximately 200 patients with Parkinson's Disease and early motor fluctuations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGI-C) score improvement (minimally, much or very much), no change or worsening (minimally, much or very much) 12 months after start of treatment. | 12 months
  To evaluate the long-term effectiveness of opicapone in patients with Parkinson's disease and early motor fluctuations by means of the PGI-C at 12 months after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Fabbrini, Principal Investigator — Azienda Universitaria Policlinico Umberto I, Roma
Locations (20):
- Italy (20):
  - Policlinico di Bari Ospedale Giovanni XXIII, Clinica Neurologia AMADUCCI, Bari
  - ASST Spedali Civili di Brescia, Brescia
  - ARNAS Azienda Ospedaliera Brotzu, Cagliari
  - Ospedale Mater Domini, Catanzaro
  - Ospedale SS Annunziata, Chieti
  - Ospedale Policlinico San Martino, Genova
  - Centro Neurolesi Bonino Pulejo Messina/IRCCS, Messina
  - ASST Gaetano Pini CTO, Centro Parkinson, Milan
  - Istituto Neurologico Carlo Besta - Fondazione IRCCS, Milan
  - U.O di Neurologia, Policlinico P. Giaccone, Palermo
  - Fondazione Mondino, Pavia
  - Azienda Ospedaliera di Perugia (Santa Maria della Misericordia), Perugia
  - Ospedale Santa Chiara, Pisa
  - Arcispedale S. Maria Nuova (AUSL RE), Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Roma
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma
  - A.O.U Città della Salute e della Scienza di Torino, Turin
  - Ospedale Borgo Roma, Verona

IPD SHARING:
Plan to Share IPD: No